CLINICAL TRIAL: NCT02180672
Title: Utility of Nasal Steroids for Treatment of Childhood Obstructive Sleep Apnea
Brief Title: Steroids for Pediatric Apnea Research in Kids
Acronym: SPARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-010942; R01HL120909 (NIH)
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive sleep apnea syndrome; OSA; sleep apnea; nasal steroids; corticosteroids
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal steroids (Active Comparator): Participants randomly assigned to this study arm will receive a 3-month course of nasal steroids (nasal fluticasone).
  Interventions: Drug: Nasal Fluticasone
- Placebo (Placebo Comparator): Participants randomly assigned to this study arm will receive a 3-month course of placebo nasal spray (saline).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nasal Fluticasone — One spray per nostril, per day.
  Other Names: NCS; Nasal steroids; Nasal corticosteroids
  Arms: Nasal steroids
Drug: Placebo — One spray per nostril, per day.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This double-blind, randomized controlled trial will evaluate the use of nasal corticosteroids for the treatment of the childhood obstructive sleep apnea syndrome (OSAS). Efficacy, duration of action and side-effects will be determined.

DETAILED DESCRIPTION:
Several studies have suggested that Nasal corticosteroids (NCS) or leukotriene antagonists may be effective in the treatment of childhood OSAS. However, these studies have been limited by factors such as small size, lack of randomization and blinding, short-term follow-up, involvement of children with only very mild OSAS, and/or lack of stratifying for the presence of atopy. Therefore, investigators will plan a randomized controlled trial evaluating the efficacy and safety of NCS vs placebo in children with mild to moderate OSAS. The overall hypothesis is that NCS will be safe and efficacious in the treatment of mild to moderate childhood OSAS, particularly in children with asthma/atopy, but will require ongoing maintenance therapy.

ELIGIBILITY:
Inclusion Criteria

1. 5-10 years of age.
2. Mild to moderate OSAS, defined as an obstructive apnea index of 1-20/hr of total sleep time or obstructive apnea hypopnea index of 2-30/hr of total sleep time.
3. Parent-related symptoms of habitual snoring (>3 nights per week)
4. No history of adenotonsillectomy.
5. Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria

1. Severe OSAS or significant hypoxemia or hypercapnia on polysomnography, such that definitive treatment should not be delayed (AHI > 30/hr, more than 2% total sleep time with arterial oxygen saturation (SpO2) <90%, end-tidal carbon dioxide partial pressure (PCO2) > 60 mm Hg for > 5 minutes, pathologic arrhythmias).
2. History of recurrent throat infections (as defined by the American Academy of Otolaryngology-Head and Neck Surgery Clinical Practice Guidelines For Tonsillectomy (7)) in the past few years as follows: > 7 episodes in the past year or > 5 episodes/year over the past 2 years or > 3 episodes/year over the past 3 years.
3. Abnormalities on baseline safety screening tests, i.e., Dual Energy X-ray Absorptiometry (DXA) scan showing spine or whole body bone mineral density < -2.0 standard deviations using race specific curves with adjustment for height Z-score; morning cortisol < 3 µg/dl or morning adrenocorticotropic hormone (ACTH) < 10 pg/ml; or ophthalmologic exam demonstrating cataracts (except those with < 2 mm anterior polar cataracts), aphakia or other ocular abnormalities such as glaucoma, retinal coloboma, intraocular inflammation or microphthalmia.
4. Failure to thrive (weight/height < 5th percentile for age and gender), as this may be secondary to OSAS.
5. Severe obesity (BMI z-score > 3) as OSAS is likely to persist in these subjects.
6. Previous adenoidectomy unless adenoidal tissue has been documented to have regrown.
7. Previous tonsillectomy.
8. Continuous positive airway pressure (CPAP) therapy.
9. Any NCS use in the past 3 months or NCS use for > 2 weeks in the past year.
10. Current immunotherapy or daily antihistamine use.
11. Recent (past month) nasal septum ulcers, surgery or trauma.
12. Other major illness other than asthma, such as craniofacial anomalies, endocrine or neuromuscular disease, or past history of cancer. This includes children with conditions that may be worsened by OSAS, such as hypertension or diabetes.
13. Current use of ketoconazole or other potent CYP3A4 inhibitors.
14. Families planning to move out of the area within the year.
15. Subjects who do not speak either English or Spanish well enough to complete the validated neurobehavioral instruments.
16. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12-30 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole L Marcus, MBBCh, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chidambaram AG, Cielo CM, Chervoneva I, Spergel JM, Tapia IE. Nasal biomarker inflammatory profile in response to intranasal corticosteroids in pediatric obstructive sleep apnea syndrome. J Clin Sleep Med. 2025 Jun 1;21(6):1033-1040. doi: 10.5664/jcsm.11604. PMID 40051199
- [Derived] Tapia IE, Shults J, Cielo CM, Kelly AB, Elden LM, Spergel JM, Bradford RM, Cornaglia MA, Sterni LM, Radcliffe J. A Trial of Intranasal Corticosteroids to Treat Childhood OSA Syndrome. Chest. 2022 Oct;162(4):899-919. doi: 10.1016/j.chest.2022.06.026. Epub 2022 Jun 30. PMID 35779610
- See also: Related Info — http://www.research.chop.edu/research/clinical-research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening: polysomnography, ophthalmologic exam, DXA scan. 75 children did not meet PSG inclusion criteria, 1 child had a coloboma, and 1 child had abnormal DXA scan.
Period: Overall Study
Arm/Group | Nasal Steroids | Placebo
Started | 91 | 43
Completed | 86 | 36
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Steroids | Placebo | Total
Number analyzed (Participants) | 91 | 43 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.24 (2.17) | 8.10 (2.03) | 8.17 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 20 | 65
  Male | 46 | 23 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 25 | 90
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 91 | 43 | 134
OAHI [Mean (Full Range); unit: events per hour] — Obstructive apnea hypopnea index (events per hour). Per inclusion/exclusion criteria the expected range for this study at baseline is between 2 and 30 events per hour. Please note that lower and upper ranges can be broader at the 3- and 12-month points. Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  events per hour
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 7.85 [6.50 to 9.20] | 6.51 [5.09 to 7.94] | 7.52 [3.40 to 9.49]
Nasal Obstrction Symptoms Evaluation (NOSE) [Mean (Full Range); unit: units on a scale] — Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated scale of nasal obstructive symptoms, modified by deleting the question about sleep and written in child-friendly language. Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  units on a scale
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 5.59 [4.60 to 6.59] | 4.47 [3.07 to 5.88] | 5.03 [3.84 to 6.24]
The Epworth Sleepiness Scale [Mean (Full Range); unit: units on a scale] — Epworth Sleepiness scale is a measure of sleepiness that ranges from 0-24, with higher values indicating sleepiness Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  units on a scale
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 9.09 [8.09 to 10.1] | 7.58 [5.54 to 9.63] | 8.34 [6.82 to 9.87]
Pediatric Quality of Life (PedsQL) [Mean (Full Range); unit: units on a scale] — Pediatric Quality of Life Inventory (PedsQL) is a well-validated, generic measure of global quality of life in which scores range from 0 to 100, with higher scores indicating better quality of life Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  units on a scale
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 73.91 [69.90 to 77.930] | 78.44 [72.0 to 84.89] | 76.175 [70.95 to 81.41]
Behavior Rating Inventory of Executive Function (BRIEF) [Mean (Full Range); unit: T-Score] — Behavior Rating Inventory of Executive Function [BRIEF] Global Executive Composite T score, comprising summary measures of behavioral regulation and metacognition [with mean scores of 50 and standard deviation of 10, with higher scores indicating worse functioning] Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  T-Score
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 50.86 [47.95 to 53.77] | 47.11 [42.52 to 51.70] | 48.985 [45.235 to 52.735]
Conners Abbreviated Symptom Questionnaire [Mean (Full Range); unit: T-Score] — The Conners Abbreviated Symptom Questionnaire is a parent-rated measure of symptoms of attention problems, yielding T scores with a mean of 50 and a standard deviation of 10 (higher scores indicate worse functioning). Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  T-Score
    number analyzed (Participants) | 86 | 36 | 122
    (all) | 8.19 [6.49 to 9.88] | 5.97 [3.81 to 8.14] | 7.08 [5.15 to 9.01]
Conners Continuous Performance Test (CPT) [Mean (Full Range); unit: T-Score] — The CPT is a performance measure of sustained attention that yields T scores with a mean of 50 and a standard deviation of 10 (higher scores indicate worse functioning) Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  T-Score
    number analyzed (Participants) | 82 | 36 | 118
    (all) | 54.8 [52.83 to 56.77] | 56.1 [52.65 to 59.55] | 55.45 [52.74 to 58.16]
Purdue Peg Board [Mean (Full Range); unit: z-Score] — The Purdue Peg Board is a widely used test of fine motor coordination, yields z-scores with a mean of 0 and a standard deviation of 1, with higher scores indicating better performance. Population: The total number of analyzed is different than the total number of participants is due to participants withdrawing themselves from the study or being lost to follow up.
  z-Score
    number analyzed (Participants) | 85 | 35 | 120
    (all) | -1.06 [-1.35 to -0.78] | -1.39 [-1.83 to 0.95] | -1.225 [-1.59 to 0.085]

OUTCOME MEASURES:

1. Primary Outcome: Obstructive Apnea Hypopnea Index
Description: Efficacy measure to assess acute response to nasal steroids.
  Obstructive apnea hypopnea index (events per hour). Per inclusion/exclusion criteria the expected range for this study at baseline is between 2 and 30 events per hour. Please note that lower and upper ranges can be broader at the 3- and 12-month points.
  The obstructive apnea hypopnea index (OAHI) is the sum of obstructive apneas and hypopneas, and mixed apneas divided by the total hours of sleep. Hence, the unit used is events per hour. It ranges from 0 events per hour(meaning no obstructive apneas at all) until 400 events per hour approximately. Higher values indicate more severe obstructive sleep apnea or worse outcome.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: events per hour
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 86 | 36
events per hour | 7.69 [5.39 to 9.99] | 6.33 [4.09 to 8.58]

2. Secondary Outcome: OAHI
Description: Efficacy measure to assess duration of response to nasal steroids.
  Obstructive apnea hypopnea index (events per hour). Per inclusion/exclusion criteria the expected range for this study at baseline is between 2 and 30 events per hour. Please note that lower and upper ranges can be broader at the 3- and 12-month points.
Time Frame: 12 months
Population: The obstructive apnea hypopnea index (OAHI) is the sum of obstructive apneas and hypopneas, and mixed apneas divided by the total hours of sleep. Hence, the unit used is events per hour. It ranges from 0 events per hour(meaning no obstructive apneas at all) until 400 events per hour approximately. Higher values indicate more severe obstructive sleep apnea or worse outcome.
Measure: Mean (95% Confidence Interval); unit: events per hour
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
events per hour | 6.11 [3.97 to 8.24] | 6.27 [3.98 to 8.55]

3. Secondary Outcome: Nasal Obstruction Symptom Evaluation (NOSE)
Description: Nasal Obstruction Symptom Evaluation (NOSE) scale, a validated scale of nasal obstructive symptoms. The scales ranges from 0-100 with higher values indicating worse nasal obstruction
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
score on a scale | 3.66 [2.54 to 4.77] | 5.31 [3.43 to 7.2]

4. Secondary Outcome: The Epworth Sleepiness Scale
Description: Epworth Sleepiness scale is a measure of sleepiness that ranges from 0-24, with higher values indicating sleepiness
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
score on a scale | 7.68 [6.24 to 9.12] | 8.56 [6.68 to 10.45]

5. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL)
Description: Pediatric Quality of Life Inventory (PedsQL), a well-validated, generic measure of global quality of life, in which scores range from 0 to 100, with higher scores indicating better quality of life
Time Frame: 12 month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
score on a scale | 78.69 [72.93 to 84.45] | 73.67 [66.66 to 80.68]

6. Secondary Outcome: Behavior Rating Inventory of Executive Function (BRIEF)
Description: Behavior Rating Inventory of Executive Function [BRIEF] Global Executive Composite T score, comprising summary measures of behavioral regulation and metacognition [with mean scores of 50 and standard deviation of 10, with higher scores indicating worse functioning]
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
T-Score | 47.42 [43.93 to 50.91] | 49.5 [44.01 to 54.99]

7. Secondary Outcome: Conners Abbreviated Symptom Questionnaire
Description: A parent-rated measure of symptoms of attention problems, yielding T scores with a mean of 50 and a standard deviation of 10 (higher scores indicate worse functioning).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 36 | 32
T-Score | 5.62 [3.73 to 7.52] | 6.50 [3.84 to 9.16]

8. Secondary Outcome: Purdue Peg Board
Description: The Purdue Peg Board is a widely used test of fine motor coordination, yields z-scores with a mean of 0 and a standard deviation of 1, with higher scores indicating better performance.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: z-Score
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 31
z-Score | -1.12 [-1.7 to -0.54] | -1.31 [-1.79 to -0.84]

9. Secondary Outcome: Conners Continuous Performance Test (CPT)
Description: The CPT is a performance measure of sustained attention that yields T scores with a mean of 50 and a standard deviation of 10 (higher scores indicate worse functioning)
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 36 | 29
T-Score | 52.67 [49.07 to 56.27] | 52.92 [48.74 to 57.11]

10. Secondary Outcome: Child Behavior Checklist
Description: The Child Behavior Checklist (CBCL), is a widely used and validated caregiver-completed survey of behavior competencies that yields standardized, age-adjusted scores on internalizing, externalizing and attentional behavior difficulties81, 82. All scores are T scores with a mean of 50 and standard deviation of 10 (higher scores indicate worse functioning).
Time Frame: 12-Months
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Nasal Steroids | Placebo
Number analyzed (Participants) | 38 | 32
T-Score
  Internalizing | 49.92 [47.01 to 52.83] | 51.94 [47.46 to 56.42]
  Externalizing | 51.89 [48.45 to 55.34] | 52 [47.34 to 56.66]
  Total Behavior Problems | 51.45 [48.47 to 54.43] | 51.19 [45.99 to 56.39]
  Attention | 55.13 [53.47 to 56.79] | 57.38 [54.15 to 60.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected monthly at telephone calls at months 2, 4, 5, 7, 8, 10 and 11, and during in-person visits at months 1, 3, 6, 9 and 12.
Arm/Group | Nasal Steroids | Placebo
All-Cause Mortality (participants affected / at risk) | 66/86 | 16/36
Serious Adverse Events (participants affected / at risk) | 1/86 | 0/36
Other Adverse Events (participants affected / at risk) | 66/86 | 16/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Steroids (N=86) | Placebo (N=36)
Ketotic Hypoglycemia (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Steroids (N=86) | Placebo (N=36)
Lower Respiratory Tract (Including Asthma) (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Upper Respiratory Tract (including cough) (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 7 (7)
Gastrointestinal Tract (Gastrointestinal disorders) | 10 (10) | 2 (2)
Other Infections (Infections and infestations) | 8 (8) | 3 (3)
Sleep Apnea Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Other Illness (General disorders) | 31 (31) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02180672/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02180672/ICF_001.pdf